CLINICAL TRIAL: NCT02756715
Title: The Effect of Anesthetics Agents on Vascular Injury and Level of Syndecan-1 During Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KUH1160100
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol group (Active Comparator): The patient who anesthetized by using propofol.
  Interventions: Drug: propofol group
- Desflurane group (Active Comparator): The patient who anesthetized by using sevoflurane.
  Interventions: Drug: Desflurane group

INTERVENTIONS:
Drug: propofol group — Patient will be anesthetized by using propofol infusion during operation.
  Other Names: Propofol
  Arms: propofol group
Drug: Desflurane group — Patient will be anesthetized by using desflurane inhalation during operation.
  Other Names: Desflurane
  Arms: Desflurane group

SUMMARY:
Ischeic reperfusion injury lead to a cellular dyfunction and increase in soluble glycocalyx of blood flow. syndecan-1 was a marker of glycocalyx.

The purpose of this study is to prove the variation of level of serum syndecan-1 between preoperative and postoperative period.

DETAILED DESCRIPTION:
The patients were allocated randomly to receive propofol or desflurane. Also, a total of 6ml of blood sample was obtained for total 6 times in consecutive order.

1. Preoperation (immediate before anesthesia induction)
2. Immediate before tourniquet off
3. 5 min after tourniquet off
4. PACU
5. postoperative 6 hours
6. postoperative 24 hours

Serum in blood will be obtained and level of serum cytokine will be evaluated by enzyme-linked immunosorbent assay

ELIGIBILITY:
Inclusion Criteria:

* patients who was planned to undergo knee surgery.

Exclusion Criteria:

* age < 20 years old
* history of previous cancer
* history of previous peripheral vascular disease
* Emergency surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Syndecan-1 | Preoperative time, Immediate before tourniquet off,5 min after tourniquet off,PACU, postoperation after 6hours, postoperation after 24hours
  change of level of syndecan-1 (scores range from 0 to 100)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D,Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh CS, Choi JM, Park EH, Piao L, Park HJ, Rhee KY, Kim SH. Impact of Anesthetic Agents on Endothelial Glycocalyx Injury during Total Knee Arthroplasty: Desflurane- vs. Propofol-Based Anesthesia-A Prospective Randomized Controlled Trial. Biomed Res Int. 2021 Jan 23;2021:8880267. doi: 10.1155/2021/8880267. eCollection 2021. PMID 33564684